CLINICAL TRIAL: NCT00757042
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 157 in Healthy Subjects and Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Safety Study of Tezepelumab (AMG 157) in Healthy Adults and Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20070620
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2022-07-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Atopic Dermatitis; Healthy Volunteers
Keywords: atopic dermatitis; skin diseases; healthy volunteer
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Escalating dose cohorts will be enrolled sequentially based on a blinded review of safety data up to day 15 of the previous dose cohort with consideration of predefined stopping rules.
  The first 2 participants in Cohort 1 will be a sentinel pair, randomized at a 1:1 ratio to receive either tezepelumab or placebo and monitored for safety and tolerability. Once the safety in the sentinel pair is confirmed the subsequent six participants will be randomized at a 5:1 ratio for tezepelumab or placebo treatment. In cohorts 2 through 8 (escalating doses, healthy subjects), participants will be randomized to receive tezepelumab or placebo at a 6:2 ratio. In cohort 9 (700 mg IV, atopic dermatitis subjects),a sentinel pair will again be used to first establish safety, and the subsequent 10 participants will be randomized to receive tezepelumab or placebo at a ratio of 8:2, for a total of 12 evaluable participants in this cohort.
Who Masked: Participant, Investigator

ARMS (2):
- Tezepelumab (Experimental): Participants will receive a single dose of tezepelumab administered subcutaneously or intravenously. The starting dose will be 2.1 mg tezepelumab.
  Interventions: Drug: Tezepelumab
- Placebo (Placebo Comparator): Participants will receive matching placebo administered subcutaneously or intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tezepelumab — Administered by subcutaneous or intravenous injection
  Other Names: AMG 157; Tezspire
  Arms: Tezepelumab
Drug: Placebo — Matching placebo administered by subcutaneous or intravenous injection.
  Arms: Placebo

SUMMARY:
This study is a single dose escalation study of tezepelumab (AMG 157) in healthy adults (Part A) and adults with moderate to severe atopic dermatitis (Part B). The purpose of the study is to evaluate the safety, tolerability, immunogenicity and pharmacokinetics of tezepelumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject must sign an Institutional Review Board (IRB) approved informed consent form before any study specific procedures
* Subjects must be aged between 18 and 45 years, inclusive (Part A only)
* Female subjects must be of non-reproductive potential
* Male subjects with partners of childbearing potential should inform their partner of their participation in this clinical study and use highly effective methods of birth control during the study
* Healthy subjects must have a body mass index (BMI) between 18 to 32 kg/m^2, inclusive
* Subject must have normal or clinically acceptable physical examination, clinical laboratory tests and electrocardiogram (ECG) results
* For Part B, subject must have active atopic dermatitis (AD) affecting ≥ 10% body surface area; Eczema Area and Severity Index (EASI) score ≥ 15, aged between 18 and 60 years, inclusive and BMI between 18 and 35 kg/m^2, inclusive

Exclusion Criteria:

* Subject who has history or evidence of a clinically significant disorder, condition or disease that, in the opinion of the Investigator in consultation with the Amgen physician, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Subject who has evidence of any active or suspected bacterial, viral, fungal or parasitic infections within the past 30 days prior to randomization
* Subject who has known positive tuberculin skin test or recent (within 6 months from randomization) exposure to an individual with active tuberculosis
* Subject who has history of malignancy within 5 years before randomization
* Subject who has history of significant dermatological conditions (except for atopic dermatitis in Part B)
* Subject who has previously received any investigational drug (or is currently using an investigational device) within 30 days prior to randomization
* Subject who has tested positive for drugs and/or alcohol use at screening or before randomization
* Female subjects who are pregnant or lactating
* Subject who has used nicotine or tobacco containing products during 6 months before randomization and during the study (except for Part B below)
* Subject has known type I/II diabetes
* Subject used nonprescription drugs within 14 days prior to randomization and during the study
* Subject used any cytotoxic or immunosuppressive drugs with 30 days or 5 half-lives prior to randomization and during the study
* Subject previously received a monoclonal antibody
* Subject donated blood or had loss of blood of equal to or greater than 500 mL with 2 months of screening
* Subject positive for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies
* Subject has any condition that might compromise informed consent or compliance to the protocol
* For atopic dermatitis subjects in Part B (Cohorts 9 and 10) only, additional exclusion criteria are as follows:
* Subject who has concurrent skin disease (eg, acne) of such severity in the study area that it could interfere with study evaluation;
* Subject who has active or recent skin infections (within 7 days of randomization);
* Subject who has received phototherapy (eg, ultraviolet [UV] A, UVB) known or suspected to have an effect on AD within 6 weeks prior to randomization;
* Subject who has received corticosteroids by other than topical, inhaled or intranasal delivery within 4 weeks prior to randomization;
* Subject who has been treated with topical calcineurin inhibitors within 14 days prior to randomization;
* Subject who uses any medications that interfere with blood coagulation (eg nonsteroidal anti-inflammatory drugs [NSAIDs]) or wound healing within 7 days or 5 half-lives (whichever is longer) prior to enrolling into the study and for the duration of the study.
* Subject who smokes more than 10 cigarettes per day within the 6 months prior to randomization and during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2008-09-18 (Actual); Primary Completion 2011-01-05 (Actual); Study Completion 2011-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Parnes JR, Sullivan JT, Chen L, Dias C. Pharmacokinetics, Safety, and Tolerability of Tezepelumab (AMG 157) in Healthy and Atopic Dermatitis Adult Subjects. Clin Pharmacol Ther. 2019 Aug;106(2):441-449. doi: 10.1002/cpt.1401. Epub 2019 Mar 23. PMID 30779339
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a single-ascending dose (SAD) study of tezepelumab in healthy adults (Part A; Cohorts 1-8) and adults with moderate to severe atopic dermatitis (AD) (Part B; Cohort 9).
  The study was conducted at seven centers in the United States, including one center that conducted the testing in all healthy adults and six centers that performed the study in AD participants.
  Dose escalation was based on blinded review of safety data up to day 15 from the previous cohort.
Pre-assignment Details: In Part A the first 2 participants enrolled in Cohort 1 were randomized in a 1:1 ratio and subsequent participants in this cohort were randomized in a 5:1 ratio to receive tezepelumab or placebo. For Cohorts 2 to 8 in Part A, participants were randomized in a 6:2 ratio to receive tezepelumab or placebo. In Part B, the first 2 participants were randomized in a 1:1 ratio, and subsequent participants in Cohort 9 were randomized in an 8:2 ratio to receive tezepelumab or placebo.
Groups:
- Part A: Tezepelumab 2.1 mg SC: Healthy participants received a single dose of 2.1 mg tezepelumab administered subcutaneously (SC).
- Part A: Tezepelumab 7 mg SC: Healthy participants received a single dose of 7 mg tezepelumab administered subcutaneously.
- Part A: Tezepelumab 21 mg SC: Healthy participants received a single dose of 21 mg tezepelumab administered subcutaneously.
- Part A: Tezepelumab 70 mg SC: Healthy participants received a single dose of 70 mg tezepelumab administered subcutaneously.
- Part A: Tezepelumab 210 mg SC: Healthy participants received a single dose of 210 mg tezepelumab administered subcutaneously.
- Part A: Tezepelumab 420 mg SC: Healthy participants received a single dose of 420 mg tezepelumab administered subcutaneously.
- Part A: Tezepelumab 210 mg IV: Healthy participants received a single dose of 210 mg tezepelumab administered intravenously.
- Part A: Tezepelumab 700 mg IV: Healthy participants received a single dose of 700 mg tezepelumab administered intravenously.
- Part A: Placebo: Healthy participants received a single dose of placebo to tezepelumab administered subcutaneously or intravenously.
- Part B: Tezepelumab 700 mg IV: Participants with atopic dermatitis received a single dose of 700 mg tezepelumab administered intravenously.
- Part B: Placebo IV: Participants with atopic dermatitis received a single dose of placebo to tezepelumab administered intravenously.
Period: Overall Study
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV | Part A: Placebo | Part B: Tezepelumab 700 mg IV | Part B: Placebo IV
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 10 | 4
Received Study Drug | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 9 | 3
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Ineligibility Determined | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of Investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV | Part A: Placebo | Part B: Tezepelumab 700 mg IV | Part B: Placebo IV | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 9 | 3 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (4.9) | 32.2 (2.1) | 36.8 (2.6) | 28.3 (4.9) | 33.7 (4.1) | 37.0 (3.7) | 33.0 (7.5) | 30.2 (3.6) | 32.3 (7.6) | 48.1 (11.3) | 45.3 (5.5) | 34.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 16
  Male | 5 | 4 | 1 | 5 | 6 | 6 | 5 | 5 | 13 | 7 | 3 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 0 | 2 | 3 | 2 | 2 | 2 | 4 | 8 | 2 | 27
  Black or African American | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 7
  Hispanic or Latino | 3 | 5 | 5 | 4 | 2 | 2 | 4 | 1 | 11 | 0 | 0 | 37
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) include any untoward medical occurrence in a trial participant administered a study drug and does not necessarily have a causal relationship with this treatment. AEs include worsening of a pre-existing medical condition and laboratory value changes requiring therapy or adjustment in prior therapy.
  AEs were assessed for severity according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3, where Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = severe AE, Grade 4 = life-threatening AE and Grade 5 = death due to AE.
  Relationship to study treatment was determined by the investigator.
  A serious adverse event (SAE) is defined as an AE that met 1 or more of below criteria:
  * was fatal;
  * was life threatening;
  * required in-patient hospitalization or prolongation of existing hospitalization;
  * resulted in persistent or significant disability/incapacity;
  * was a congenital anomaly/birth defect;
  * other significant medical hazard.
Time Frame: For Part A Tezepelumab/Placebo 2.1 mg, 7 mg, 21 mg, 70 mg, and 210 mg SC: 85 days. For Part A Tezepelumab/Placebo 420 mg SC, 210 mg IV, and 700 mg IV and Part B: 113 days
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo SC: Healthy participants received a single dose of placebo to tezepelumab administered subcutaneously.
- Part A: Placebo IV: Healthy participants received a single dose of placebo to tezepelumab administered intravenously.
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV | Part A: Placebo SC | Part A: Placebo IV | Part B: Tezepelumab 700 mg IV | Part B: Placebo IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 9 | 3
Participants
  Any adverse event | 3 | 5 | 1 | 6 | 2 | 3 | 4 | 5 | 8 | 3 | 7 | 3
  Serious adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AE leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to discontinuation from study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse event | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 4 | 1 | 3 | 3

2. Secondary Outcome: Part A: Time of Maximum Observed Concentration (Tmax) of Tezepelumab
Description: The time at which the maximum concentration of tezepelumab was observed was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The concentration of tezepelumab in human serum was measured using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: Day 1 predose, 0.25, 0.5, and 1 hour after start of infusion (for IV cohorts only), 4, 8, 24, 48, 72 hours postdose and days 5, 6, 7, 11, 15, 22, 29, 43, 57, 71, 85, and (for cohorts who received 420 mg tezepelumab SC or any IV dose) 113.
Population: Participants in Part A who received tezepelumab and had a sufficient number of serum concentration measurements for computing the pharmacokinetic (PK) parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 190.94 [117.87 to 332.15] | 237.09 [140.50 to 335.07] | 142.10 [117.43 to 336.10] | 130.87 [69.27 to 237.90] | 93.65 [70.22 to 359.17] | 80.89 [68.27 to 116.58] | 1.13 [1.08 to 8.00] | 1.04 [1.02 to 1.17]

3. Primary Outcome: Number of Participants Who Developed Anti-tezepelumab Antibodies
Description: All study samples (tezepelumab and placebo) were tested using an electrochemiluminescence (ECL) based immunoassay to detect and confirm the presence of antibodies capable of binding to tezepelumab. Samples identified as positive in the immunoassay were tested in a receptor-binding ECL-based assay to detect neutralizing or inhibitory effects toward tezepelumab.
  The number of participants with positive anti-tezepelumab binding antibodies / neutralizing antibodies at any time post-baseline with a negative or no result at baseline is reported.
Time Frame: Blood samples for the measurement of antibodies were collected on Days 29, 57, 85, and (for cohorts who received 420 mg Tezepelumab/placebo SC or any IV dose) 113.
Population: All participants who received at least 1 dose of study drug with a postbaseline result.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV | Part A: Placebo | Part B: Tezepelumab 700 mg IV | Part B: Placebo IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 15 | 9 | 3
Participants
  Anti-tezepelumab binding antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Anti-tezepelumab neutralizing antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) of Tezepelumab
Description: The maximum observed serum concentration of tezepelumab was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The concentration of tezepelumab in human serum was measured using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: as for outcome 2
Population: Participants in Part A who received tezepelumab and had a sufficient number of serum concentration measurements for computing the PK parameter.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
μg/mL | 0.257 (0.0824) | 0.792 (0.0593) | 2.01 (0.620) | 7.82 (2.25) | 23.6 (10.3) | 58.0 (19.3) | 64.4 (10.2) | 219 (38.3)

5. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Tezepelumab
Description: The PK parameter AUC0-t was estimated based on the serum concentrations of tezepelumab using noncompartmental methods and the linear/log trapezoidal method. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
day*μg/mL | 8.12 (1.96) | 32.9 (2.75) | 76.7 (31.6) | 278 (64.3) | 867 (349) | 2050 (627) | 1150 (176) | 3440 (253)

6. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of Tezepelumab
Description: The PK parameter AUCinf was estimated based on the serum concentrations of tezepelumab using noncompartmental methods and the linear/log trapezoidal method. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
day*μg/mL | 8.69 (1.97) | 36.6 (4.60) | 84.6 (37.9) | 303 (70.3) | 976 (409) | 2140 (677) | 1200 (208) | 3530 (322)

7. Secondary Outcome: Part A: Elimination Half-life (t1/2) of Tezepelumab
Description: Elimination half-life was estimated based on the serum concentrations of tezepelumab using noncompartmental methods based on the terminal phase of the concentration-time profile.
  The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
days | 19.9 (4.81) | 23.4 (4.30) | 22.7 (4.81) | 22.5 (1.35) | 25.7 (5.52) | 23.3 (2.89) | 24.5 (6.28) | 20.7 (6.44)

8. Secondary Outcome: Part B: Time of Maximum Observed Concentration (Tmax) of Tezepelumab
Description: Tmax was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: Day 1 predose, 0.25, 0.5, 1, 4, 8, 72 hours postdose and days, 7, 15, 22, 29, 43, 57, 71, 85, and 113.
Population: Participants in Part B who received tezepelumab and had a sufficient number of serum concentration measurements for computing the PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Part B: Tezepelumab 700 mg IV
Number analyzed (Participants) | 9
hours | 4.08 [1.00 to 8.12]

9. Secondary Outcome: Part B: Maximum Observed Concentration (Cmax) of Tezepelumab
Description: Cmax was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: Day 1 predose, 0.25, 0.5, 1, 4, 8, 72 hours postdose and days, 7, 15, 22, 29, 43, 57, 71, 85, and 113.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part B: Tezepelumab 700 mg IV
Number analyzed (Participants) | 9
μg/mL | 253 (57.2)

10. Secondary Outcome: Part B: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Tezepelumab
Description: as for outcome 5
Time Frame: Day 1 predose, 0.25, 0.5, 1, 4, 8, 72 hours postdose and days, 7, 15, 22, 29, 43, 57, 71, 85, and 113.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Part B: Tezepelumab 700 mg IV
Number analyzed (Participants) | 9
day*μg/mL | 3660 (990)

11. Secondary Outcome: Part B: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of Tezepelumab
Description: as for outcome 6
Time Frame: Day 1 predose, 0.25, 0.5, 1, 4, 8, 72 hours postdose and days, 7, 15, 22, 29, 43, 57, 71, 85, and 113.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Part B: Tezepelumab 700 mg IV
Number analyzed (Participants) | 9
day*μg/mL | 3830 (1230)

12. Secondary Outcome: Part B: Elimination Half-life (t1/2) of Tezepelumab
Description: as for outcome 7
Time Frame: Day 1 predose, 0.25, 0.5, 1, 4, 8, 72 hours postdose and days, 7, 15, 22, 29, 43, 57, 71, 85, and 113.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part B: Tezepelumab 700 mg IV
Number analyzed (Participants) | 9
days | 22.2 (4.72)

13. Secondary Outcome: Part B: Percentage of Participants Achieving at Least a 50% Reduction From Baseline in Eczema Area and Severity Index (EASI 50) Score
Description: EASI is a tool used to measure the severity of AD. The index involves an assessment of the average intensity of 4 clinical signs (erythema, infiltration/papulation, excoriations, and lichenification) at 4 body areas (head/neck, upper extremities, trunk, lower extremities) assessed on a scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe.
  The percent of affected area for each of the 4 body areas is also assessed using the following 6-point scale: 0 = 0%, 1 = < 10%, 2 =10% to 29%, 3 = 30% to 49%, 4 = 50% to 69%, 5 = 70% to 89%, 6 = 90% to 100%. The total score for each body region is obtained by multiplying the sum of the severity scores of the 4 clinical signs by the area score, with adjustment for the proportion of the body region to the whole body.
  The sum of the scores for each body region gives the total EASI score, which ranges from 0 to 72, with higher scores indicating greater disease severity.
Time Frame: Baseline and days 15, 29, 43, 57, 85, and 113
Population: All participants in Part B who received at least 1 dose of study drug and with available data at each time point.
Measure: Number; unit: percentage of participants
Groups:
- Part B: Placebo: Participants with atopic dermatitis received a single dose of placebo to tezepelumab administered intravenously.
Arm/Group | Part B: Tezepelumab 700 mg IV | Part B: Placebo
Number analyzed (Participants) | 9 | 3
percentage of participants
  Day 15 | 22 | 0
  Day 29 | 22 | 0
  Day 43 | 22 | 33
  Day 57: number analyzed (Participants) | 9 | 2
  Day 57 | 22 | 0
  Day 85: number analyzed (Participants) | 8 | 3
  Day 85 | 50 | 0
  Day 113 | 33 | 33
  At any postdose time point | 56 | 33

14. Secondary Outcome: Part B: Percentage of Participants Achieving at Least a 75% Reduction From Baseline in Eczema Area and Severity Index (EASI 75) Score
Description: as for outcome 13
Time Frame: Baseline and days 15, 29, 43, 57, 85, and 113
Population: All participants in Part B who received at least 1 dose of study drug and with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tezepelumab 700 mg IV | Part B: Placebo
Number analyzed (Participants) | 9 | 3
percentage of participants
  Day 15 | 0 | 0
  Day 29 | 0 | 0
  Day 43 | 0 | 0
  Day 57: number analyzed (Participants) | 9 | 2
  Day 57 | 11 | 0
  Day 85: number analyzed (Participants) | 8 | 3
  Day 85 | 13 | 0
  Day 113 | 22 | 0
  At any postdose time point | 22 | 0

15. Secondary Outcome: Part B: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: EASI is a tool used to measure the severity of AD. The index involves an assessment of the intensity of 4 clinical signs (erythema, infiltration/papulation, excoriations, and lichenification) at 4 body areas (head/neck, upper extremities, trunk, lower extremities) assessed on a scale from 0 (none) to 3 (severe).
  The percent affected area for each of the 4 body areas is assessed on a 6-point scale from 0 (0%) to 6 (90% to 100%). The total score for each body region is obtained by multiplying the sum of the severity scores of the 4 clinical signs by the area score, with adjustment for the proportion of the body region to the whole body.
  The total EASI score is the sum of the scores for each body region, and ranges from 0 to 72, with higher scores indicating greater disease severity.
  Percent change from baseline = [(Post-baseline Value - Baseline Value) / Baseline Value] x 100.
  A negative change from baseline indicates improvement.
Time Frame: Baseline and days 15, 29, 43, 57, 85, and 113
Population: All participants in Part B who received at least 1 dose of study drug and with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part B: Tezepelumab 700 mg IV | Part B: Placebo
Number analyzed (Participants) | 9 | 3
percent change
  Day 15 | -12.47 (43.32) | 15.10 (55.84)
  Day 29 | -23.61 (32.82) | -25.03 (20.38)
  Day 43 | -17.04 (44.28) | -32.41 (31.81)
  Day 57: number analyzed (Participants) | 9 | 2
  Day 57 | -22.83 (41.23) | -1.89 (37.24)
  Day 85: number analyzed (Participants) | 8 | 3
  Day 85 | -31.70 (42.14) | -23.01 (21.16)
  Day 113 | -25.25 (49.40) | -11.28 (54.63)

16. Secondary Outcome: Part B: Change From Baseline in Investigator's Global Assessment (IGA)
Description: IGA score is a static 6-point measure of disease activity based on an overall assessment of skin lesions. The IGA was scored on a scale of 0 to 5, where 0 (clear) = no inflammatory signs of AD;
  1. (almost clear) = just perceptible erythema and just perceptible papulation/infiltration;
  2. (mild) = mild erythema and mild papulation and infiltration;
  3. (moderate) = moderate erythema and moderate papulation and infiltration;
  4. (severe) = severe disease with severe erythema and severe papulation and infiltration;
  5. (very severe) = severe disease with severe erythema and severe papulation and infiltration with oozing/crusting.
  A negative change from baseline indicates improvement.
Time Frame: Baseline and days 15, 29, 43, 57, 85, and 113
Population: All participants in Part B who received at least 1 dose of study drug and with available data at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part B: Tezepelumab 700 mg IV | Part B: Placebo
Number analyzed (Participants) | 9 | 3
scores on a scale
  Day 15 | -0.33 (0.50) | 0.33 (0.58)
  Day 29 | -0.56 (0.73) | -0.67 (0.58)
  Day 43 | -0.44 (0.53) | -1.00 (0.00)
  Day 57: number analyzed (Participants) | 9 | 2
  Day 57 | -0.44 (0.73) | -1.00 (0.00)
  Day 85: number analyzed (Participants) | 8 | 3
  Day 85 | -0.63 (0.74) | -1.33 (0.58)
  Day 113 | -0.44 (0.73) | -0.33 (1.15)

ADVERSE EVENTS:
Time Frame: For Part A Tezepelumab/Placebo 2.1 mg, 7 mg, 21 mg, 70 mg, and 210 mg SC: 85 days. For Part A Tezepelumab/Placebo 420 mg SC, 210 mg IV, and 700 mg IV and Part B: 113 days
Arm/Group | Part A: Tezepelumab 2.1 mg SC | Part A: Tezepelumab 7 mg SC | Part A: Tezepelumab 21 mg SC | Part A: Tezepelumab 70 mg SC | Part A: Tezepelumab 210 mg SC | Part A: Tezepelumab 420 mg SC | Part A: Tezepelumab 210 mg IV | Part A: Tezepelumab 700 mg IV | Part A: Placebo SC | Part A: Placebo IV | Part B: Tezepelumab 700 mg IV | Part B: Placebo IV
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/4 | 0/9 | 1/3
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 1/6 | 6/6 | 2/6 | 3/6 | 4/6 | 5/6 | 8/12 | 3/4 | 7/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Tezepelumab 2.1 mg SC (N=6) | Part A: Tezepelumab 7 mg SC (N=6) | Part A: Tezepelumab 21 mg SC (N=6) | Part A: Tezepelumab 70 mg SC (N=6) | Part A: Tezepelumab 210 mg SC (N=6) | Part A: Tezepelumab 420 mg SC (N=6) | Part A: Tezepelumab 210 mg IV (N=6) | Part A: Tezepelumab 700 mg IV (N=6) | Part A: Placebo SC (N=12) | Part A: Placebo IV (N=4) | Part B: Tezepelumab 700 mg IV (N=9) | Part B: Placebo IV (N=3)
INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Tezepelumab 2.1 mg SC (N=6) | Part A: Tezepelumab 7 mg SC (N=6) | Part A: Tezepelumab 21 mg SC (N=6) | Part A: Tezepelumab 70 mg SC (N=6) | Part A: Tezepelumab 210 mg SC (N=6) | Part A: Tezepelumab 420 mg SC (N=6) | Part A: Tezepelumab 210 mg IV (N=6) | Part A: Tezepelumab 700 mg IV (N=6) | Part A: Placebo SC (N=12) | Part A: Placebo IV (N=4) | Part B: Tezepelumab 700 mg IV (N=9) | Part B: Placebo IV (N=3)
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
KERATITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
APPLICATION SITE URTICARIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
INJECTION SITE HAEMORRHAGE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HAEMATOMA INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TINEA CRURIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 4 | 1 | 2 | 1
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEPATIC ENZYME ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
LIBIDO DECREASED (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.